CLINICAL TRIAL: NCT05918874
Title: Evaluation of Postnatal Nutritional Status and Physical Activity Level in Obese Asthmatic Children
Brief Title: Postnatal Nutrition and Physical Activity in Obese Asthmatic Children
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozden Gokcek, Principal Investigator, Ege University
Other Study IDs: 2023/15
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Asthma in Children
Keywords: Childhood asthma; Obesity; Physical activity; Postnatal nutrition
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese: The demographic characteristics of the children, type of asthma, dietary habits, socioeconomic income level and number of meals were asked to the child; the use of vitamin D in childhood and for how long, whether the child was breastfed or not, how many months the child was breastfed if breastfed, whether the mother had a smoking habit, and whether the mother had urinary tract infection during pregnancy were asked to the mother.
  Asthma control level was recorded according to the asthma control test. Body mass index was calculated according to the Center of Disease Control and Prevention. The leisure-time activity scale and the International Physical Activity Questionnaire for Children-C (IPAQ-C) were used to assess physical activity level.
  Interventions: Other: Descriptive questionnaire
- non-obese: The demographic characteristics of the children, type of asthma, dietary habits, socioeconomic income level and number of meals were asked to the child; the use of vitamin D in childhood and for how long, whether the child was breastfed or not, how many months the child was breastfed if breastfed, whether the mother had a smoking habit, and whether the mother had urinary tract infection during pregnancy were asked to the mother.
  Asthma control level was recorded according to the asthma control test. Body mass index was calculated according to the Center of Disease Control and Prevention. The leisure-time activity scale and the International Physical Activity Questionnaire for Children-C (IPAQ-C) were used to assess physical activity level.
  Interventions: Other: Descriptive questionnaire

INTERVENTIONS:
Other: Descriptive questionnaire — Questionnaires were administered to calculate whether the children were obese or not, to determine their asthma control levels, to determine their physical activity levels and to determine their leisure time activities.

SUMMARY:
The aim of this study was to compare the duration of breast milk intake, vitamin D intake, asthma control level and physical activity levels between obese asthmatic children and non-obese children. This was a prospective study in children aged 8-17 years with asthma. Asthma control level was evaluated by asthma control test and physical activity level was evaluated by Physical Activity Questionnaire for Children (IPAQ-C) and leisure time activity scale.

DETAILED DESCRIPTION:
Asthma and obesity, which are important public health problems and are common in childhood, are chronic diseases. The aim of this study was to compare breastfeeding duration, vitamin D intake, asthma control and physical activity levels between obese asthmatic children and non-obese children.

The study was a prospective study conducted in children aged 8-17 years with asthma. Demographic information of the children was recorded. Asthma control level was assessed by asthma control test and physical activity level was assessed by Physical Activity Questionnaire for Children (IPAQ-C) and leisure time activity scale.

It was conducted as a single-blind, prospective study in which the patients were randomized by simple randomization method as obese asthmatic children (experimental group) and non-obese asthmatic children (control group) according to the order of admission to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with asthma by a pediatrician,
* not in the attack process,
* no mental problems,
* do not have any systemic disease accompanying asthma (diabetes, etc.)
* children who voluntarily agreed to participate in the study

Exclusion Criteria:

* severe posture disorders
* idiopathic scoliosis and idiopathic rheumatic disease
* history of orthopedic surgery
* children with mental retardation or a neurological problem

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Volunteer children between the ages of 8-17 years with a diagnosis of asthma admitted to the Department of Pediatrics.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-01-23 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 4 months
  Percentages were calculated with the CDC (Center of Disease Control and Prevention) BMI Percentage Calculator for Children and Adolescents.
Sedentary time spent by children | 4 months
  Children's Leisure Time Activity Survey (CLASS)
Physical activity levels of children | 4 months
  International Physical Activity Questionnaire for Children (IPAQ-C)

SECONDARY OUTCOMES:
Asthma control level | 4 months
  Asthma Control Test
Demographic information questionnaire | 4 months
  The child was asked about demographic characteristics, asthma type, dietary habits, socioeconomic income level and number of meals; the mother was asked whether she used vitamin D during childhood and for how long; whether the child received breast milk and if so, for how many months; whether the mother had a smoking habit; and whether the mother had a urinary tract infection during pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege university faculty of health sciences, Izmir, Karsıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data sets generated and/or analyzed during the current study may be made available from the relevant principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF